CLINICAL TRIAL: NCT04726878
Title: Effectiveness of the Erector Spinae Plane Block in Patients Undergoing Breast Surgery Due to Cancer
Brief Title: ESP in Breast Surgery Due to Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Michał Borys, associate professor, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KE-0254/92/2018
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Pain, Acute; Anesthesia, Local
Keywords: erector spinae plane block; visual analog scale; quality of recovery; patient-controlled analgesia
MeSH Terms: conditions — Breast Neoplasms; Acute Pain | interventions — Anesthesia, General; Analgesia, Patient-Controlled; Passive Cutaneous Anaphylaxis; Oxycodone; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1:1
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient: The primary intervention (erector spinae plane block) will be provided under general anesthesia.
  The investigator and outcome assessor will be not aware of the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controlled (Placebo Comparator): Standard care without regional block. General anesthesia. After the end of the surgery, the patient-controlled analgesia with oxycodone.
  Interventions: Procedure: General anesthesia; Procedure: Patient-controlled analgesia; Drug: Oxycodone; Drug: paracetamol
- ESP block (Experimental): After the induction of general anesthesia, before the beginning of the surgery, the erector spinae plane block with 0.375% ropivacaine will be performed. Then, the patient will be treated as in the controlled group.
  Interventions: Procedure: Erector spinae plane block; Procedure: General anesthesia; Procedure: Patient-controlled analgesia; Drug: Oxycodone; Drug: paracetamol
- Sham block (Sham Comparator): After the induction of general anesthesia, before the beginning of the surgery, the erector spinae plane block with 0.9% saline will be performed. Then, the patient will be treated as in the controlled group.
  Interventions: Procedure: Sham block; Procedure: General anesthesia; Procedure: Patient-controlled analgesia; Drug: Oxycodone; Drug: paracetamol

INTERVENTIONS:
Procedure: Erector spinae plane block — Ultrasound-guided the erector spinae plane block with 0.375% ropivacaine, 0.4 mL per KG, up to 40 mL (maximum dose).
  Other Names: ESP block
  Arms: ESP block
Procedure: Sham block — Ultrasound-guided the erector spinae plane block with 0.9% saline, 0.4 mL per KG, up to 40 mL (maximum dose).
  Arms: Sham block
Procedure: General anesthesia — Standard general anesthesia. The induction with fentanyl, 1-3 mcg per KG; propofol, 1.5-2 mg per kg. Then, the laryngeal mask airway will be inserted. Patients with the risk of aspiration will be intubated using rocuronium or suxamethonium.
  The maintenance with oxygen/air mixture, sevoflurane, and fentanyl.
  Other Names: GA
Procedure: Patient-controlled analgesia — All patients will receive a PCA pump with oxycodone (1 mg/mL, 5-minute interval) after transfer to PACU (post-anesthesia care unit)
  Other Names: PCA
Drug: Oxycodone — Intravenous oxycodone will be administered about 30 minutes before the end of the surgery at a dose of 0.1 mg/KG. Additional 2 doses can be given if pain on the visual analog scale will be higher than 40.
Drug: paracetamol — intravenous paracetamol will be used (1.0 gram), up to 4 grams per day

SUMMARY:
Patients scheduled for breast surgery due to cancer. Each patient will be treated with intravenous (i.v.) oxycodone - patient-controlled analgesia (PCA). Patients will be allocated to one of three groups: erector spinae plane (ESP) block, sham block, controlled group.

DETAILED DESCRIPTION:
Only patients who are qualified for an elective procedure of mitral breast surgery may participate in the study. Each patient will be anesthetized generally. The same drugs will be used in each stage of anesthesia. The induction: propofol, fentanyl, rocuronium. The airway will be secured with a laryngeal mask airway (LMA). When there is a risk of aspiration, the patient will be intubated. Then, rocuronium or suxamethonium will be used. The anesthesia maintenance: sevoflurane, fentanyl. The emergence: oxygen, sugammadex or neostigmine a required.

After the induction of general anesthesia, an opaque envelope with the selected group will be opened. In the controlled group, the procedure will be continued in the patient's supine position. Women from the ESP and Sham groups will be placed in the lateral position. The operated side will be above. Then, the ultrasound-guided ESP block with saline or ropivacaine will be performed.

At the end of the surgery, an anesthesiologist will administer oxycodone intravenously (0.1 mg/KG).

After emergence from anesthesia, the patient will be transferred to the postoperative care unit. Vital signs will be monitored. The patient-controlled analgesia pump with oxycodone will be used.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery of breast due to cancer
* obtained consent

Exclusion Criteria:

* the lack of consent
* the surgery of two breasts
* reoperation of the same breast
* previous participation in the study
* coagulopathy
* allergy to morphine and local anesthetics
* depression, antidepressant drugs treatment
* epilepsy
* usage of painkiller before surgery
* addiction to alcohol or recreational drugs

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Quality of recovery 40 | Before the hospital discharge
  Quality of recovery (QoR) score containing 40 items. This questionnaire measures the early postoperative health status of patients. Minimum is 40, maximum is 200. More points is better.

SECONDARY OUTCOMES:
Patient-controlled analgesia (PCA) | 24 hours from the connection of the PCA pump in the post-anesthesia care unit.
  All good and bad demands with PCA pump.
Visual analog scale | up to 24 hours after the surgery
  Acute pain measured with VAS (visual analog scale). From 0 (no pain) to 100. More on the scale is worse.
Total oxycodone consumption | up to 24 hours after the surgery
  Consumption of oxycodone with PCA pump, loading, and additional doses.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Piwowarczyk, MD-PhD, Study Chair — Medical University of Lublin
Locations (1):
- II Department of Anesthesia and Intensive Care, Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiech M, Piwowarczyk P, Mieszkowski M, Tuyakov B, Pituch-Sala K, Czarnik T, Kurylcio A, Czuczwar M, Borys M. The quality of recovery after erector spinae plane block in patients undergoing breast surgery: a randomized controlled trial. BMC Anesthesiol. 2022 Jul 14;22(1):222. doi: 10.1186/s12871-022-01760-z. PMID 35836116